CLINICAL TRIAL: NCT05202535
Title: Effect of Aerobic Exercise Training on Arterial Stiffness and Hemodynamics in Obese Adults.
Brief Title: Effect of Aerobic Exercise Training in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01092 Khowla shah
Record Dates: First submitted 2022-01-08; First posted 2022-01-21 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Obesity
Keywords: Aerobic exercise, arterial stiffness, hemodynamics, obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise training (Experimental): hospital-based aerobic exercise training on treadmill/cycle ergometer with the intensity of 40-70% of HR max, for 15-30 mints for 8 weeks
  Interventions: Other: Aerobic exercise training
- Conventional therapy (Active Comparator): Patient education and counseling with diet plan.Walking 3 days15min/day for 8 weeks
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Aerobic exercise training — Hospital-based aerobic exercise training for 15-30 minutes including pre and post-vitals assessment.
  3x/week on alternate days for 8 weeks at 40-70% of HR Max
  Arms: Aerobic exercise training
Other: Conventional therapy — Patient education and counseling with diet plan.Walking 3 days15min/day for 8 weeks
  Arms: Conventional therapy

SUMMARY:
To determine the effect of aerobic exercise training on arterial stiffness and hemodynamics in obese adults. Proper evidence on the effect of aerobic exercise training on both arterial stiffness and hemodynamics are sparsely present in obese adults whereas separate studies were done in mainly hypertensive and cardiovascular disease populations.

DETAILED DESCRIPTION:
Obese adults always have been trying to improve their quality of life by managing the complications associated with obesity like arterial stiffness and disturbed hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥28 kg/m²
* Able to do exercise

Exclusion Criteria:

* Involved in structured physical activity in last 6 months
* History of chronic systemic disease (cardiovascular, pulmonary, and metabolic disease)
* Continuous medication use.
* MSK or Neurological problems
* Pregnant females

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Arterial Stiffness | 6 weeks
  Gradual fragmentation and loss of elastin fibers and accumulation of stiffer collagen fibers in the arterial wall. Calculated through Arterial stiffness index.
Hemodynamics | 6 weeks
  Factors that govern blood flow calculated through Rate Pressure Product.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Polyclinic Hospital, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hvidt KN. Blood pressure and arterial stiffness in obese children and adolescents. Dan Med J. 2015 Mar;62(3):B5043. PMID 25748874
- [Background] Cote AT, Phillips AA, Harris KC, Sandor GG, Panagiotopoulos C, Devlin AM. Obesity and arterial stiffness in children: systematic review and meta-analysis. Arterioscler Thromb Vasc Biol. 2015 Apr;35(4):1038-44. doi: 10.1161/ATVBAHA.114.305062. Epub 2015 Jan 29. PMID 25633314